CLINICAL TRIAL: NCT05708794
Title: A Pilot Study to Assess Feasibility of Evaluating the Safety and Efficiency of a Simplified Diagnostic Approach for Pulmonary Embolism
Brief Title: Adjust-Unlikely PE
Status: Completed | Type: Observational
Sponsor: Dr. Kerstin de Wit (Other)
Collaborators: Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network)
Responsible Party: Sponsor-Investigator, Dr. Kerstin de Wit, Dr. Kerstin de Wit, Associate Professor, Department of Emergency Medicine, Queen's University, Queen's University
Organization: Queen's University (Other)
Other Study IDs: 4269
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Embolism (Diagnosis)
Keywords: emergency medicine; standardization of practice; diagnostics evaluation
MeSH Terms: conditions — Pulmonary Embolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this pilot study is to assess the feasibility of a larger study to determine the Adjust-Unlikely algorithm safety and efficiency for diagnosing PE.

The pilot study objectives are to:

1. Determine study recruitment rate, per site, per month
2. Determine study 90-day loss to follow up rate
3. Estimate of the proportion of enrolled patients who test negative for PE at initial assessment using the Adjust-Unlikely rule
4. Estimate of the Adjust-Unlikely algorithm efficiency
5. Compare excluded and missed-eligible patients to study participants: age, sex and prevalence of PE diagnoses at initial testing.

The pilot study hypothesis is that the investigators can recruit at least 20 patients per month and successfully follow at least 90% of patients for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Emergency physician decides to test for PE

Exclusion Criteria:

* Tested for PE without using the Adjust-Unlikely algorithm
* D-dimer level is known before Adjust-Unlikely assessment
* A new indication for anticoagulation on emergency department assessment (other than pulmonary embolism) in a patient not previously prescribed an anticoagulant
* Declines participation
* Is inaccessible for follow-up
* Has previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to emergency departments and urgent care centres with symptoms of PE.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who have PE excluded by the Adjust-Unlikely algorithm and who are subsequently diagnosed with either PE or lower limb DVT. | 90 days following index presentation

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin de Wit, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No